CLINICAL TRIAL: NCT02791724
Title: Evaluating a Novel Cognitive-Behavioral Online Depression Intervention for Persons With Epilepsy (Desiconnect): Randomized Controlled Trial
Brief Title: Evaluating a Novel Internet Intervention for Persons With Epilepsy and Depression
Acronym: ENCODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EP28b_01
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Depression; Epilepsy
MeSH Terms: conditions — Depression; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desiconnect (Experimental): Desiconnect is an Internet-administered intervention developed for persons with epilepsy and elevated depression symptoms.
  Interventions: Behavioral: Desiconnect; Other: CAU
- Care-as-Usual (CAU) / wait list (Active Comparator): In the CAU/wait list control group, participants are free to continue to engage with any treatment they require (i.e., CAU). However, they will receive access to Desiconnect three months post-baseline (i.e., wait list with respect to Desiconnect access).
  Interventions: Other: CAU

INTERVENTIONS:
Behavioral: Desiconnect — Desiconnect is an Internet intervention for persons with epilepsy and elevated depression. Content is continuously adapted to patients' concerns and needs. Techniques to overcome depression (e.g., cognitive restructuring, behavioral activation) and to cope with anxiety symptoms (e.g., exposure, role of avoidance, mindfulness exercises) are conveyed in interactive sequences that are accompanied by audio recordings, illustrations, and worksheets. Topics covered also include coping with epilepsy symptoms, identifying and coping with seizure auras and triggers, and the role of nutrition and exercise. Patients are also prompted to regularly complete brief symptom severity self-monitoring questionnaires. Optional daily text messages with motivational content accompany the program. The program can be accessed for 180 days after registration.
  Arms: Desiconnect
Other: CAU — Care as Usual

SUMMARY:
The trial aims to evaluate the effectiveness of a novel internet intervention (Desiconnect), which was designed to introduce relevant cognitive-behavioral therapy (CBT) techniques to Persons with Epilepsy (PwE) and comorbid depression. Therefore, 200 PwE and a current depressive disorder (major depressive disorder or dysthymic disorder) will be recruited and randomized to two groups: (1) a control group, in which they may engage with any epilepsy treatment (Care-as-Usual, CAU) and receive access to Desiconnect after a delay of three months (i.e., CAU/wait list control group), or (2) to a treatment group that immediately receives six-month access to Desiconnect and may also use CAU. The primary outcome measure is the depression scale of the Patient Health Questionnaire (PHQ-9), collected at three months post-baseline.

DETAILED DESCRIPTION:
Depression is common among persons with epilepsy (PwE), affecting roughly one in three individuals, and its presence is associated with personal suffering, impaired quality of life, and worse prognosis. Despite the availability of effective treatments, depression is often overlooked and treated inadequately in PwE, in part because of concerns over drug interactions. Previous studies strongly suggest that cognitive behavioral therapy (CBT) can help alleviate depression in PwE, but CBT is not always available to patients. Internet-administered psychological interventions are easily accessible and might complement antidepressant medication or psychotherapy, and preliminary evidence suggests that such interventions can be effective. However, no trial has yet examined whether a CBT-based internet intervention designed to meet the needs of PwE can achieve sustained reductions in depression and related symptoms, such as anxiety, when offered as adjunct to treatment as usual.

The Internet-based intervention evaluated in this trial was designed with the aim of conveying evidence-based psychotherapeutic techniques, gleaned primarily from CBT, to PwE over a period of 180 days. The intervention focuses on identifying and challenging cognitions that trigger or sustain depression and anxiety, increasing activities that are likely to reduce depression and anxiety, practicing relaxation and stress management exercises and increasing mindfulness skills. The program is based on general CBT and other evidence-based psychotherapeutic techniques that have been shown to be helpful for patients suffering from depression (and ideally, that have been shown to be helpful among PwE). Furthermore, program content addresses other issues in disease self-management, including lifestyle habits (e.g., nutrition, exercise) and medication adherence. The delivery and training of content is continuously individualized to match users' preferences and needs, based on responses within the program. The intervention is delivered via the Internet and protected by individually assigned passwords.

This randomized controlled trial will include 200 participants with epilepsy and a current depressive disorder, along with currently at least moderately elevated depression. Participants will be recruited from various settings, including epilepsy treatment clinics, outpatient treatment centers, and Internet forums/groups. Methods such as newspaper articles, flyers, posters, and media articles or web-advertisements will be used to inform potential participants about the study (all material will be in German). Participants will be randomly assigned to either (1) a control group, in which they receive care as usual (CAU) and are given access to the internet intervention (Desiconnect) after a delay of 3 months (i.e., CAU/Wait list control group), or (2) a treatment group that may also use CAU and in addition immediately receives six-month access to the novel, internet-administered intervention (Desiconnect). Measurements are collected online at pre-treatment (baseline, T0), three months (T1), six months (T2), and nine months (T3).

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* diagnosis of active epilepsy (that is, at least one epileptic seizure within the past 10 years or taking antiseizure medicines within the past five years)
* current depressive disorder (either major depressive disorder or dysthymic disorder, as determined by telephone interview with the MINI Neuropsychiatric Interview)
* no current antidepressant medication, or current antidepressant medication but no changes in dosage for at least one month prior to study inclusion (medication changes after study inclusion are permitted, given the pragmatic design of the trial)
* currently at least moderate self-reported depressive symptom severity, as operationalized by a score of at least 10 on the PHQ-9, a cut-off score that has been well validated
* ability to speak and read German
* access to the internet and personal possession of an appropriate device on which the internet-based intervention can be used regularly (e.g., smartphone, computer, laptop)
* expressed motivation to participate in the trial and use an internet-based intervention to acquire skills and knowledge that may aid in the amelioration of depression symptoms

Exclusion Criteria:

* current psychotherapy
* other known major psychiatric disorder, such as bipolar disorder, schizophrenia or another psychotic disorder, or borderline personality disorder (based on the MINI interview)
* acute suicidality (that is, intention or plan to commit suicide, as assessed with the respective module of the MINI interview)
* newly prescribed antidepressant medication or change in antidepressant medication dosage in month prior to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptoms, measured by Patient Health Questionnaire - 9 items (PHQ-9) | Change from baseline to 3 months (also assessed at 6 and 9 months post-baseline)
  Self-report depression symptom severity measure

SECONDARY OUTCOMES:
NDDIE (Neurological Disorders Depression Inventory for Epilepsy) | Change from baseline to 3 months (also assessed at 6 and 9 months post-baseline)
  Epilepsy-specific self-report measure of depression symptom severity
GAD-7 (Generalized Anxiety Disorder Questionnaire) | Change from baseline to 3 months (also assessed at 6 and 9 months post-baseline)
  Self-report anxiety symptom severity measure
DASS-21 (Depression and Anxiety Scales) | Change from baseline to 3 months (also assessed at 6 and 9 months post-baseline)
  Self-report measure of anxiety, depression, and stress symptoms
WSAS (Work and Social Adjustment Scale) | Change from baseline to 3 months (also assessed at 6 and 9 months post-baseline)
  Self-report measure of depression-related psychosocial impairment
Subjective usefulness of the program | Assessed at 3 and 6 months
  Individually designed self-report items
INEP (Inventory for the Assessment of Negative Effects of Psychotherapy) | Assessed at 3 and 6 months
  Adapted self-report measure assessing potential negative effects of the Internet intervention
PESOS | Assessed at baseline, 3, 6, and 9 months
  Self-report measure of epilepsy symptoms
LSSS (Liverpool Seizure Severity Scale) | Assessed at baseline, 3, 6, and 9 months
  Self-report measure of epilepsy symptoms
QOLIE-10 (Health-related Quality of Life) | Assessed at baseline, 3, 6, and 9 months
  Self-report measure of health-related quality of life
ESMS (Epilepsy Self-Management Scale) | Assessed at baseline, 3, 6, and 9 months
  Self-report measure of epilepsy self-management practices

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Ph.D., Principal Investigator — University Medical Center Hamburg-Eppendorf (UKE), Department of Psychosomatic Medicine and Psychotherapy
Locations (1):
- University Medical Center Hamburg-Eppendorf (UKE), Department of Psychiatry and Psychotherapy, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data shall be made available upon request for projects such as meta-analyses after completion of the study

REFERENCES:
- [Background] Meyer B, Weiss M, Holtkamp M, Arnold S, Bruckner K, Schroder J, Scheibe F, Nestoriuc Y. Protocol for the ENCODE trial: evaluating a novel online depression intervention for persons with epilepsy. BMC Psychiatry. 2017 Feb 7;17(1):55. doi: 10.1186/s12888-017-1229-y. PMID 28173780
- [Result] Meyer B, Weiss M, Holtkamp M, Arnold S, Bruckner K, Schroder J, Scheibe F, Nestoriuc Y. Effects of an epilepsy-specific Internet intervention (Emyna) on depression: Results of the ENCODE randomized controlled trial. Epilepsia. 2019 Apr;60(4):656-668. doi: 10.1111/epi.14673. Epub 2019 Feb 25. PMID 30802941